CLINICAL TRIAL: NCT02226588
Title: Two Community Strategies Comparing Use of Misoprostol for Secondary Prevention to Primary Prevention for Postpartum Hemorrhage: A Randomized Cluster Non-Inferiority Study in El Beheira Governorate, Egypt
Brief Title: Comparison of Primary and Secondary Prevention of Postpartum Hemorrhage at the Community Level in Egypt
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Ministry of Health and Population, Egypt (Other Government); University of Alexandria (Other); El Galaa Teaching Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3004
Record Dates: First submitted 2014-08-25; First posted 2014-08-27 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Secondary prevention (Experimental): Single sublingual dose of 800mcg (4 tablets) misoprostol administered to women with 350-500mL postpartum blood loss as estimated using a blood absorption mat or due to deteriorating postpartum condition of the woman as determined by provider's clinical judgment
  Interventions: Drug: Misoprostol
- Universal prophylaxis (Active Comparator): Single oral prophylactic dose of 600mcg (3 tablets) misoprostol administered to all women within 1 minute of deliver of baby
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol

SUMMARY:
The objective of this study is to compare two community-level strategies: either selective, early administration of 800 mcg sublingual misoprostol to women for secondary prevention of postpartum hemorrhage (PPH) or universal use of 600 mcg oral misoprostol at the time of delivery for prophylaxis of PPH. The significance of this cluster randomized non-inferiority trial is its potential to inform service delivery programs on clinical outcomes, program feasibility, cost, and acceptability of two different community models of PPH care using misoprostol.1. The study hypothesizes that a service delivery model that administers misoprostol for secondary prevention is non-inferior to a model that administers misoprostol for universal prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent
* Vaginal delivery
* Agrees to participate in follow-up interview
* Agrees to have pre- and post-hemoglobin taken
* Delivery at woman's home or at the primary health unit (PHU)

Exclusion Criteria:

* Too advanced into active labor to provide consent
* Known allergy to misoprostol and/or other prostaglandin
* Pregnancy complications, such as hypertension, suspected multiple pregnancy, previous caesarean section, suspected still birth, ante-partum hemorrhage, and previous complication in the third trimester

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2827 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Mean drop in pre- to post-delivery hemoglobin level | Pre-delivery hemoglobin will be measured during a third trimester antenatal care visit or during early labor. Post-delivery hemoglbin will be measured 2 to 4 days after delivery of the baby.
  Hemoglobin will be measured by primary health unit staff using a portable handheld Hemocue machine.

SECONDARY OUTCOMES:
Proportion of women transferred to higher level care | Following delivery to postpartum visit (2 to 4 days after delivery)
  The proportion of women transferred to higher level care will be assessed. Includes the condition of woman at time of transfer and arrival at transfer facility.
Proportion of women diagnosed with PPH | After delivery of the baby up to 24 hours postpartum
  PPH will be diagnosed using the standard practices of PHU staff
Proportion of women receiving additional interventions for PPH | Following delivery to postpartum visit (2 to 4 days after delivery)
  An additional intervention could include: uterotonics, manual removal of placental fragments. bimanual compression, IV fluids given to control active bleeding.
Proportion of women who experience side effects | From time of delivery to 2 hours postpartum
  Women experiencing known side effects of misoprostol, including shivering/chills and pyrexia; severity, duration, and any additional care provided will be assessed
Proportion of women who find the intervention acceptable | Measured at postpartum visit (2 to 4 days after delivery)
  Acceptability will be assessed in an exit interview with women - women will be asked if they are willing to take misoprostol in future deliveries and about the preferences what method they would prefer (primary or secondary prevention) in future deliveries.
Proportion of women who receive intervention per protocol | within 2 hours of delivery
  To assess feasibility, we will document the proportion of women for whom the intervention arm protocol is correctly followed (including correct timing of drug administration, when necessary).
Proportion of women experiencing a serious adverse event | Within 2 to 4 days after delivery
  Serious adverse events include hysterectomy, blood transfusion, maternal death

CONTACTS AND LOCATIONS:
Overall Officials: Nevine Hassanein, MD, Principal Investigator — Consultant; Emad Darwish, MD, Principal Investigator — Alexandria University; Mohamed Cherine, MD, Principal Investigator — El Galaa Teaching Hospital; Rasha Dabash, MPH, Principal Investigator — Gynuity Health Projects; Holly Anger, MPH, Principal Investigator — Gynuity Health Projects
Locations (2):
- Egypt (2):
  - Primary Health Care Units, Damanhur, El Beheira
  - Primary Health Care Units, Kafr El Dawar, El Beheira

REFERENCES:
- [Derived] Anger HA, Dabash R, Hassanein N, Darwish E, Ramadan MC, Nawar M, Charles D, Breebaart M, Winikoff B. A cluster-randomized, non-inferiority trial comparing use of misoprostol for universal prophylaxis vs. secondary prevention of postpartum hemorrhage among community level births in Egypt. BMC Pregnancy Childbirth. 2020 May 24;20(1):317. doi: 10.1186/s12884-020-03008-5. PMID 32448257
- See also: Related Info — http://www.gynuity.org